CLINICAL TRIAL: NCT00560547
Title: An Open Label Study to Assess the Maintenance of Hemoglobin Levels, Safety and Tolerability of Once Monthly Administration of Mircera in Hemodialysis Patients With Chronic Renal Anemia.
Brief Title: A Study of Once-Monthly Intravenous Mircera in Hemodialysis Patients With Chronic Renal Anemia.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was cancelled before any patients were enrolled, due to operational reasons.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21349
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — 120, 200 or 360 micrograms / 4 weeks iv (starting dose)
  Other Names: Mircera

SUMMARY:
This single arm study will assess the long-term maintenance of hemoglobin levels, safety and tolerability of once-monthly intravenous administration of Mircera in hemodialysis patients with chronic renal anemia. Patients currently receiving darboepoetin alfa or epoetin alfa maintenance treatment will receive intravenous Mircera at a starting dose of 120, 200 or 360 micrograms/4 weeks (based on the ESA dose administered on week-1). Subsequent doses will be adjusted to maintain hemoglobin levels within the target range of 10.5-12.5g/dL. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* regular long-term hemodialysis therapy with the same mode of dialysis for >=3 months;
* continuous iv or sc maintenance ESA treatment during previous 2 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* significant acute or chronic bleeding, such as overt gastrointestinal bleeding;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients maintaining average Hb concentration within target range during evaluation period | Weeks 17-24

SECONDARY OUTCOMES:
Change in Hb concentration between reference and evaluation period; mean time spent in, and percentage of patients maintaining Hb within target range | Weeks 17-24
Dose adjustments; RBC transfusions | Throughout study
AEs, laboratory parameters, vital signs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Denmark (3):
  - Aalborg
  - Fredericia
  - Roskilde